CLINICAL TRIAL: NCT01307683
Title: Maternal, Adiposity, Metabolism, and Stress Study (MAMAS)
Brief Title: Maternal, Adiposity, Metabolism, and Stress Study
Acronym: MAMAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: California Pacific Medical Center Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1U01HL097973 (NIH)
Record Dates: First submitted 2011-01-19; First posted 2011-03-03 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Obesity; Gestational Weight Gain
Keywords: Pregnancy; Overweight; Obese; Stress; Mindfulness
MeSH Terms: conditions — Obesity; Gestational Weight Gain; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindful Moms (Active Comparator): Based on the Mindful Motherhood Training (developed by Cassandra Vieten, PhD), Mindfulness-Based-Eating and Awareness Training (MB-EAT) (developed by Jean Kristeller, PhD), and other mindfulness- and acceptance-based interventions
  Interventions: Behavioral: Mindful Moms
- Comparison Group (No Intervention): Usual prenatal care

INTERVENTIONS:
Behavioral: Mindful Moms — 8 weekly 2-hour sessions, 2 "booster" telephone sessions, and 1 postpartum "booster" session
  Arms: Mindful Moms

SUMMARY:
The MAMAS study is built on the premise that simple recommendations for diet and exercise may not be enough to encourage healthy weight gain during pregnancy. Psychological skills training may be necessary to help women deal with stress and cravings; learn to regulate difficult emotions; increase awareness; and encourage healthy eating and physical activity. The goal of this study is to find out whether a behavioral stress reduction intervention can help women achieve healthy weight gain during pregnancy and reduce stress.

DETAILED DESCRIPTION:
The MAMAS study is adapting and testing interventions - "Moms in Joy," based on Emotional Brain Training (EBT) (developed by Laurel Mellin) and "Mindful Moms," (MIND) based on the Mindful Motherhood Training (developed by Cassandra Vieten, PhD), Mindfulness-Based-Eating and Awareness Training (MB-EAT) (developed by Jean Kristeller, PhD), and other mindfulness- and acceptance-based interventions.

In the first phase of this study, the investigators conducted in-depth focus groups with over 60 overweight, low to middle-income, pregnant women to learn more about what they might be looking for in such an intervention. In the second phase, which began in fall 2010, 48 low- to middle-income overweight pregnant women were randomly assigned to one of the interventions. Based on the knowledge gained from Phase 2, we refined the MIND intervention and are conducting an efficacy trial in Phase 3.

During Phase 3, we will enroll 220 overweight, low to middle-income, pregnant women in a trial of MIND to test feasibility and to examine changes in hypothesized mechanisms (stress, opioid tone), non-homeostatic eating, and in health outcomes (abdominal fat, insulin sensitivity, weight change) in the intervention group (n=110). Intervention participants will complete a battery of psychological and clinical measures (weight, BMI, waist/hip ratio, body composition) at baseline, post-intervention, 32-34 weeks gestation, and 3 and 9 months postpartum. Control participants (n=110) will complete the same battery of psychological measures at baseline and 8-10 weeks after baseline. All study participants will complete brief psychological, weight and waist/hip ratio measures at 6 months postpartum. Additionally, we will obtain prenatal and labor/delivery medical records for all study participants.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Currently pregnant, target 8-19 weeks gestation (intervention starts at 12-19 weeks gestation)
* Singleton gestation
* Age 18 to 45 years
* Pre-pregnancy BMI 25-41 and < 300 pounds
* Income to poverty ratio ≤ 500% specific to family size

Exclusion Criteria:

* Inability to provide informed consent or speak English (intervention is in English)
* Needle phobic or fainting in response to blood draw
* Substance abuse, mental health, or medical condition that, in the opinion of investigators, will make it difficult for the potential participant to participate in the group intervention and/or affects baseline metabolism or body composition (e.g., hypertension, asthma, arthritis, severe food allergies, HIV).
* Eating disorder which would make it difficult for the potential participant to follow the exercise, diet, and mind-body training guidelines.
* Polycystic ovarian syndrome treated with Metformin since this is indicative of insulin resistance and makes long term weight loss difficult, which are relevant outcomes in this study
* Diabetes or positive early diabetes screening test in the current pregnancy (weight loss is affected by insulin resistance)
* Previous or current mindfulness meditation practice with a typically sitting meditation of 20 or more minutes two or more times per week
* Recent weight loss (more than 5% within past 6 months). In addition, women with a history of known coronary artery disease (CAD), or typical or atypical anginal chest pain will require a letter from the participant's physician that he or she has been adequately evaluated and that a moderate exercise program is appropriate. A study physician must review the case and agree. Study participation involves a moderate exercise program. Although moderate exercise is recommended for persons with CAD, we want to ensure that steps have been taken to limit the risks of the exercise component.
* Chronic use of systemic (oral or IV) corticosteroids in the 6 months prior to enrollment (steroid use may reduce the efficacy of the intervention)
* History of gastric bypass surgery
* Multiple gestation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Adequacy of gestational weight gain, as determined by Institute of Medicine guidelines | Duration of pregnancy
  For weight change, difference between weight at the last prenatal visit before delivery, and pre-pregnancy was calculated, and categorized as inadequate, adequate and excessive weight gain according to IOM categories.

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Epel, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University California San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Epel E, Laraia B, Coleman-Phox K, Leung C, Vieten C, Mellin L, Kristeller JL, Thomas M, Stotland N, Bush N, Lustig RH, Dallman M, Hecht FM, Adler N. Effects of a Mindfulness-Based Intervention on Distress, Weight Gain, and Glucose Control for Pregnant Low-Income Women: A Quasi-Experimental Trial Using the ORBIT Model. Int J Behav Med. 2019 Oct;26(5):461-473. doi: 10.1007/s12529-019-09779-2. PMID 30993601
- [Derived] Roubinov DS, Epel ES, Coccia M, Coleman-Phox K, Vieten C, Adler NE, Laraia B, Bush NR. Long-term effects of a prenatal mindfulness intervention on depressive symptoms in a diverse sample of women. J Consult Clin Psychol. 2022 Dec;90(12):942-949. doi: 10.1037/ccp0000776. Epub 2022 Nov 28. PMID 36441994
- [Derived] Parikh NI, Laria B, Nah G, Singhal M, Vittinghoff E, Vieten C, Stotland N, Coleman-Phox K, Adler N, Albert MA, Epel E. Cardiovascular Disease-Related Pregnancy Complications Are Associated with Increased Maternal Levels and Trajectories of Cardiovascular Disease Biomarkers During and After Pregnancy. J Womens Health (Larchmt). 2020 Oct;29(10):1283-1291. doi: 10.1089/jwh.2018.7560. Epub 2020 Jan 14. PMID 31934809
- [Derived] Vieten C, Laraia BA, Kristeller J, Adler N, Coleman-Phox K, Bush NR, Wahbeh H, Duncan LG, Epel E. The mindful moms training: development of a mindfulness-based intervention to reduce stress and overeating during pregnancy. BMC Pregnancy Childbirth. 2018 Jun 1;18(1):201. doi: 10.1186/s12884-018-1757-6. PMID 29859038
- See also: University of California, San Francisco Center for Obesity Assessment, Study and Treatment — http://www.chc.ucsf.edu/coast/